CLINICAL TRIAL: NCT03162263
Title: Does Ekso Improve Motor Function and Neuroplasticity in Pazients Affected by Chronic Stroke? A Rondomized Pilot Study
Brief Title: Improving Functional Outcomes and Neuroplasticity by Using Ekso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Principal investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43/2016
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2017-08

CONDITIONS: Stroke
Keywords: Ekso; neuroplasticity; functional recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ekso training (Experimental): All patients underwent twenty-four Ekso sessions, scheduled 3 times a week. Each session lasted about 1h, and included transferring into the device arranged on an office chair; donning, standing, walking, sitting, doffing; and transferring out of the exoskeleton.The user can stand up, sit down, and walk with help of a front-wheeled walker and with the exoskeleton attached to a ceiling rail tether. A physical therapist initially provides assistance to maintain the user's center of mass over the base of support to prevent falling.
  Interventions: Device: EKso training
- Overground training (Active Comparator): Conventional gait training overground; before the training 10 min lower limb muscular exercises and stretching were performed by the physiotherapist. The overground training had the same duration of the Ekso training.
  Interventions: Device: EKso training

INTERVENTIONS:
Device: EKso training — Patients affected by chronic stroke underwent gait training by using the Ekso device; they performed a total of 20 sessions (5 day/week for 4 weeks) of at leat 40min duration.

SUMMARY:
The use of neurorobotic devices into gait rehabilitative programs, including Ekso, is reported to increase the engagement and motivation of the patients while actively performing a task, and to shape the sensory-motor plasticity (SMP) and its balance between the primary motor areas (M1), and the fronto-parietal network (FPN) connectivity, thus contributing to successful gait rehabilitation. Aim of our study was to assess whether Ekso would foster the recovery of deteriorated FPN connectivity and SMP patterns involved in limb coordination during walking in a sample of patients with hemiparesis due to stroke.

Twenty outpatients were consecutively included in this study according to the following inclusion criteria: (i) age ≥55 years; (ii) a first-ever ischemic supra-tentorial stroke (confirmed by MRI scan) at least 6 months before their enrollment; (iii) an unilateral hemiparesis, with a Muscle Research Council -MCR- score ≤3; (iv) ability to follow verbal instructions, with a Mini-Mental State Examination (MMSE) >24; (v) a Modified Ashworth Scale (MAS) score ≤2; (vi) no severe bone or joint disease; and (vii) no history of concomitant neurodegenerative diseases or brain surgery.

Patients were randomly assigned to the experimental (Ekso gait training -EGT) of control group (conventional overground gait training -OGT- at a velocity matched to the Ekso gait training).

DETAILED DESCRIPTION:
Ekso (Ekso Bionics; Richmond -CA- USA) is a wearable robot consisting of an exoskeleton framework for the lower limbs with (1) electric motors to power movement for the hip and knee joints, (2) passive spring-loaded ankle joints, (3) foot plates on which the user stands, and (4) a backpack that houses a computer, battery supply, and wired controller. A rigid backpack is an integral structural component of the exoskeleton, which provides support from the posterior pelvis to the upper back, besides carrying the computer and batteries. The exoskeleton attaches to the user's body with straps over the dorsum of the foot, anterior shin and thigh, abdomen, and anterior shoulders. The limb and pelvic segments are adjustable to the user's leg and thigh length, and the segment across the pelvis is adjustable for hip width and hip abduction angle. We preliminarily measured M1-leg excitability and SMI, which were probed using TMS pulses with a monophasic pulse configuration and peripheral nerve electric stimuli. Single magnetic pulses were given to the affected and unaffected leg-M1 using a standard figure-of-eight coil (diameter of each wing, 90 mm) connected with a high-power Magstim200 stimulator (Magstim Co, Ltd; UK).

Effective connectivity (that measures the causal influence that one brain area exerts over another under the assumption of a given mechanistic model) was assessed using a structural equation modelling (SEM). An 8-channel wireless surface EMG (sEMG) device (BTS; Milan, Italy) was used to record EMG activity from eight muscles (both tibialis anterior -TA-, soleus -S-, rectus femoris -RF-, and biceps femoris -BF). The device was also equipped with an accelerometer, put at lumbar level, to establish gait phases. Gait analysis was conducted on a 10-meter walkway.

We measured the following gait measures for both the affected and unaffected lower limb [20]: (i) step cadence (number of steps per minute; normal values 1.9±0.1 Hz);. (ii) gait cycle duration (time from one right heel strike -initial contact- to the next one -end of terminal swing; normal values 1.1±0.1 sec); (iii) stance/swing ratio (ratio between stance from heel strike to toe-off, and swing phase duration from toe-off to heel strike; normal values 1.5±0.1); .and (iv) an overall gait performance score (gait index, reflecting an approximate 60:40% distribution of stance:swing phases; normal values >90).

ELIGIBILITY:
Inclusion Criteria:

(i) age ≥55 years; (ii) a first-ever ischemic supra-tentorial stroke (confirmed by MRI scan) at least 6 months before their enrollment; (iii) an unilateral hemiparesis, with a Muscle Research Council -MCR- score ≤3; (iv) ability to follow verbal instructions, with a Mini-Mental State Examination (MMSE) >24; (v) a Modified Ashworth Scale (MAS) score ≤2; (vi) no severe bone or joint disease; and (vii) no history of concomitant neurodegenerative diseases or brain surgery.

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Motricity Index | Six months
  a measure to evaluate lower limb motor function

SECONDARY OUTCOMES:
Frontoparietotemporal connettivity | Six months
  an EEG evaluation of the patient's plasticity

CONTACTS AND LOCATIONS:
Overall Officials: Placido Bramanti, MD, Study Chair — IRCCS Neurolesi
Locations (1):
- IRCCS Centro Neurolesi Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calabro RS, Naro A, Russo M, Bramanti P, Carioti L, Balletta T, Buda A, Manuli A, Filoni S, Bramanti A. Shaping neuroplasticity by using powered exoskeletons in patients with stroke: a randomized clinical trial. J Neuroeng Rehabil. 2018 Apr 25;15(1):35. doi: 10.1186/s12984-018-0377-8. PMID 29695280